CLINICAL TRIAL: NCT04457687
Title: Extended Access Program and Retrospective Chart Review for Lorcaserin in Dravet Syndrome and Other Refractory Epilepsies
Brief Title: Extended Access Program With Lorcaserin For The Treatment of Dravet Syndrome and Other Refractory Epilepsies
Status: Available | Type: Expanded Access
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: E2023-A001-405
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Epilepsies, Myoclonic; Drug Resistant Epilepsy
Keywords: Extended Access Program; Expanded Access Program; Dravet Syndrome; Refractory Epilepsies; Lorcaserin
MeSH Terms: conditions — Epilepsies, Myoclonic; Drug Resistant Epilepsy | interventions — lorcaserin

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Lorcaserin — Lorcaserin 10 milligram (mg) tablets orally.
  Other Names: E2023

SUMMARY:
The primary purpose of this study is to provide continued access of lorcaserin to participants with Dravet syndrome and other refractory epilepsies.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of Dravet syndrome (according to Recommendation from a North American Consensus Panel, 2017) or other refractory epilepsy (per the judgment of the treating physician)
2. Male or female, age at least 2 years at the time of informed consent
3. Currently treated with lorcaserin, that the treatment is for Dravet syndrome or other refractory epilepsies, and the treatment was initiated before 13 Feb 2020; or has completed Study E2023-A001-304
4. Has a clinical benefit from lorcaserin in the opinion of the treating physician

Exclusion Criteria:

None

Min Age: 2 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (22):
- United States (18):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - David Geffen School of Medicine, UCLA Mattel Children's Hospital, Los Angeles, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Pena, Avon, Connecticut
  - (Resor), Greenwich, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Clinical Neurosciences of Tampa Bay, Clearwater, Florida
  - Miami Children's Hospital - Nicklaus Children's Hospital Miami, Miami, Florida
  - Mid-Atlantic Epilepsy and Sleep Center - Bethesda, Bethesda, Maryland
  - University of Missouri Health Care, Columbia, Missouri
  - Northeastern Regional Epilepsy Group (Hackensack), Hackensack, New Jersey
  - New York Medical College, Hawthorne, New York
  - NYU Langone Comprehensive Epilepsy Center, New York, New York
  - Mt. Sinai School of Medicine, New York, New York
  - University Hospital Cleveland Medical Center, Cleveland, Ohio
  - Sidney Kimmel Medical College at Thomas Jefferson University, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - The University of Texas Health Science Center at Houston, Houston, Texas
- Canada (4):
  - Alberta Children's Hospita, Calgary, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta
  - BC Children's Hospital, Vancouver, British Columbia
  - Children's Hospital - VH, London Health Sciences Centre, London, Ontario